CLINICAL TRIAL: NCT04124913
Title: Comparison of Oral Dydrogesterone Versus Micronized Vaginal Progesterone for Luteal Phase Support in Frozen-thawed Embryo Transfer Cycles: a Randomized Controlled Trial
Brief Title: Oral Dydrogesterone vs. Micronized Vaginal Progesterone for Luteal Phase Support in Frozen-thawed Embryo Transfer Cycles
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Memorial Sisli Hospital, Istanbul (Other)
Responsible Party: Principal Investigator, Gönül Özer, Medical doctor, Memorial Sisli Hospital, Istanbul
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2019/001
Record Dates: First submitted 2019-10-10; First posted 2019-10-14 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Infertility, Female; Infertility, Male; Embryo Transfer; Fertilization in Vitro; Drug Effect; Reproductive Techniques, Assisted; Progesterone; Dydrogesterone
Keywords: oral dydrogesterone; luteal phase support; vaginal progesterone gel; frozen-thawed embryo transfer
MeSH Terms: conditions — Infertility, Female; Infertility, Male; Helping Behavior | interventions — Dydrogesterone; Tablets; Crinone

STUDY DESIGN:
Intervention Model Description: Randomized controlled trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Dydrogesterone (Experimental)
  Interventions: Drug: Dydrogesterone 10 MG Oral Tablet
- Vaginal progesterone (Active Comparator)
  Interventions: Drug: Progesterone Vaginal Gel [Crinone]

INTERVENTIONS:
Drug: Dydrogesterone 10 MG Oral Tablet — Oral dydrogesterone 10 mg tablet three times a day for luteal phase support
  Other Names: Duphaston
  Arms: Dydrogesterone
Drug: Progesterone Vaginal Gel [Crinone] — Vaginal progesterone gel 90 mg once a day for luteal phase support
  Other Names: Crinone %8 vaginal progesterone gel
  Arms: Vaginal progesterone

SUMMARY:
The aim of this randomized controlled trial is to compare the efficacy of oral dydrogesterone vs. micronized vaginal progesterone for luteal phase support in frozen-thawed embryo transfer cycles.

ELIGIBILITY:
Inclusion Criteria:

* Ages between 20 and 40
* Modified natural frozen- thawed embryo transfer cycles

Exclusion Criteria:

* Recurrent implantation failure
* Recurrent pregnancy loss
* Presence of uterine pathology

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 140 (Estimated)
Dates: Start 2019-01-02 (Actual); Primary Completion 2019-10 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Ongoing pregnancy rate | 12 weeks after the last menstrual period of the patient
  Presence of at least one live fetus at the end of the 12th gestational week

SECONDARY OUTCOMES:
Clinical pregnancy rate | 6-7 weeks after the last menstrual period of the patient
  Presence of an intrauterine gestational sac with fetal heart beat at 7th week of gestation
Implantation rate | 5 weeks after the last menstrual period of the patient
  Percentage of gestational sacs compared to the number of embryos transferred
Biochemical pregnancy | 10 days after embryo transfer
  Positive serum beta HCG test performed 10 days after embryo transfer
Biochemical miscarriage | before 5th gestational week
  pregnancy loss before ultrasonographic detection of an intrauterine gestational sac
Clinical miscarriage | after 5th gestational week
  pregnancy loss after ultrasonographic detection of an intrauterine gestational sac
headache rate | 6-7 weeks after the last menstrual period of the patient
interference with coitus rate | 6-7 weeks after the last menstrual period of the patient
somnolence rate | 6-7 weeks after the last menstrual period of the patient
dizziness rate | 6-7 weeks after the last menstrual period of the patient
nausea/vomiting rate | 6-7 weeks after the last menstrual period of the patient
vaginal discharge rate | 6-7 weeks after the last menstrual period of the patient
perineal irritation rate | 6-7 weeks after the last menstrual period of the patient
abdominal pain rate | 6-7 weeks after the last menstrual period of the patient
mastalgia rate | 6-7 weeks after the last menstrual period of the patient
vaginal bleeding rate | 6-7 weeks after the last menstrual period of the patient
interference with intercourse rate | 6-7 weeks after the last menstrual period of the patient
overall satisfaction score | 6-7 weeks after the last menstrual period of the patient
  patient satisfaction from the drug used measured on a 1-5 scale

CONTACTS AND LOCATIONS:
Overall Officials: Semra Kahraman, Prof, Principal Investigator — Memorial Şişli Hospital
Locations (1):
- Memorial Şişli Hospital, Istanbul, Şişli, Turkey (Türkiye)